CLINICAL TRIAL: NCT01079130
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Different Doses of Indacaterol in Adult Patients With Persistent Asthma, Using Salmeterol as an Active Control
Brief Title: Efficacy and Safety of Different Doses of Indacaterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2357
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Asthma
Keywords: Indacaterol; asthma; salmeterol
MeSH Terms: conditions — Asthma | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Indacaterol 18.75 µg (Experimental): Indacaterol 18.75 µg once daily in the morning via Concept1, a single-dose dry powder inhaler (SDDPI) and Placebo to Salmeterol in the morning and in the evening via Diskus®, a multi-dose dry powder inhaler (MDDPI) for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol 37.5 µg (Experimental): Indacaterol 37.5 µg once daily in the morning via Concept1, a SDDPI and Placebo to Salmeterol in the morning and in the evening via Diskus®, a MDDPI for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol 75 µg (Experimental): Indacaterol 75 µg once daily in the morning via Concept1, a SDDPI and Placebo to Salmeterol in the morning and in the evening via Diskus®, a MDDPI for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol 150 µg (Experimental): Indacaterol 150 µg once daily in the morning via Concept1, a SDDPI and Placebo to Salmeterol in the morning and in the evening via Diskus®, MDDPI for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Salmeterol
- Salmeterol (Active Comparator): Salmeterol 50 µg twice daily in the morning and in the evening via Diskus®, a multi-dose dry powder inhaler (MDDPI) and Placebo to Indacaterol once daily in the morning via Concept1, a SDDPI for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Salmeterol; Drug: Placebo to Indacaterol
- Placebo (Placebo Comparator): Placebo to Indacaterol once daily in the morning via Concept 1, a SDDPI and Placebo to Salmeterol in the morning and in the evening via Diskus®, a MDDPI for 2 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol

INTERVENTIONS:
Drug: Indacaterol — Once daily via Concept1, a single-dose dry powder inhaler (SDDPI) for two week. Dosage varies according to randomization scheme.
  Arms: Indacaterol 150 µg; Indacaterol 18.75 µg; Indacaterol 37.5 µg; Indacaterol 75 µg
Drug: Salmeterol — 50 µg Salmeterol twice daily in the morning and in the evening via Diskus®, a MDDPI for 2 weeks.
  Arms: Salmeterol
Drug: Placebo to Indacaterol — Placebo to Indacaterol once daily in the morning via Concept 1, a SDDPI.
  Arms: Placebo; Salmeterol
Drug: Placebo to Salmeterol — Placebo to Salmeterol twice daily in the morning and in the evening via Diskus®, a multi-dose dry powder inhaler (MDDPI).
  Arms: Indacaterol 150 µg; Indacaterol 18.75 µg; Indacaterol 37.5 µg; Indacaterol 75 µg; Placebo

SUMMARY:
This study compared the 14-day bronchodilator efficacy of indacaterol with that of placebo and salmeterol

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of asthma, and:

  1. Receiving daily treatment with inhaled corticosteroid in a regimen that has been stable for at least a month prior to screening
  2. Prebronchodilator forced expiratory volume in 1 second (FEV1) at screening ≥50 and ≤90% of predicted normal
  3. An increase of ≥12% and ≥200 mL in FEV1 over prebronchodilator value within 30 minutes after inhaling albuterol

Exclusion Criteria:

* Smoking history >10 pack-years
* Patients with a diagnosis of chronic obstructive pulmonary disease (COPD)
* Patients with seasonal allergy whose asthma is likely to deteriorate during the study period
* Patients who have experienced a severe asthma attack/exacerbation requiring hospitalization in the 6 months prior to screening
* Patients who have had an intubation for a severe asthma exacerbation
* Patients who have had an emergency room visit for an asthma attack/asthma exacerbation within 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions
* Patients who have ever received or are currently receiving omalizumab or chronic oral corticosteroid therapy

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (67):
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigator Site, Scottsdale, Arizona
  - Novartis Investigator Site, Encinitas, California
  - Novartis Investigator Site, Huntington Beach, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigator Site, Orange, California
  - Novartis Investigator Site, Rancho Mirage, California
  - Novartis Investigator Site, Rolling Hills Estates, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, San Jose, California
  - Novartis Investigator Site, Stockton, California
  - Novartis Investigator Site, Colorado Springs, Colorado
  - Novartis Investigator Site, Denver, Colorado
  - Novartis Investigator Site, Engelwood, Colorado
  - Novartis Investigator Site, Lakewood, Colorado
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative site, Destin, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigator Site, Boise, Idaho
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigator Site, Overland Park, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigator Site, Lafayette, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigator Site, Columbia, Maryland
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Columbia, Missouri
  - Novartis Investigator Site, Rolla, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Warrensburg, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigator Site, Bellevue, Nebraska
  - Novartis Investigator Site, Boys Town, Nebraska
  - Novartis Investigative Site, Ocean City, New Jersey
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigator Site, Cadiz, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Maumee, Ohio
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigator Site, Portland, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Phoenixville, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Upland, Pennsylvania
  - Novartis Investigative Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative site, North Charleston, South Carolina
  - Novartis Investigator Site, Austin, Texas
  - Novartis Investigator Site, Dallas, Texas
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigator Site, Georgetown, Texas
  - Novartis Investigator Site, North Richland Hills, Texas
  - Novartis Investigator Site, Waco, Texas
  - Novartis Investigator Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 14 day run-in period. 511 participants were randomized but only 502 participants received study drug.
Period: Overall Study
Arm/Group | Indacaterol 18.75 µg | Indacaterol 37.5 µg | Indacaterol 75 µg | Indacaterol 150 µg | Salmeterol | Placebo
Started | 85 | 85 | 84 | 86 | 86 | 85
Safety Set: Received Study Drug | 84 | 81 | 84 | 85 | 84 | 84
Full Analysis Set (FAS) | 84 | 80 (2 patients (1 in 37.5 µg;1 in 75 µg group) randomized more than once and were excluded from the FAS.) | 83 | 85 | 84 | 84
Completed | 83 | 78 | 83 | 81 | 78 | 80
Not Completed | 2 | 7 | 1 | 5 | 8 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 5 | 1
Not completed — Administrative problems | 1 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 3
Not completed — Protocol deviation | 0 | 2 | 1 | 2 | 0 | 0
Not completed — Abnormal test procedure result(s) | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 18.75 µg | Indacaterol 37.5 µg | Indacaterol 75 µg | Indacaterol 150 µg | Salmeterol | Placebo | Total
Number analyzed (Participants) | 84 | 81 | 84 | 85 | 84 | 84 | 502
Age Continuous [Mean (Standard Deviation); unit: years] — All baseline measures are based on the Full Analysis Set (FAS) that includes all participants who received at least one dose of study drug.
  years | 42.0 (14.64) | 41.9 (14.96) | 40.2 (14.71) | 41.0 (15.20) | 40.9 (14.56) | 40.6 (14.17) | 41.1 (14.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 49 | 55 | 46 | 40 | 278
  Male | 42 | 35 | 35 | 30 | 38 | 44 | 224

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 2 Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. The trough FEV1 was defined as the average of the FEV1 measurements taken at 23 hours 10 minutes and 23 hours 45 minutes post dose. The mixed model used baseline FEV1 and FEV1 prior to and 30 minutes post inhalation of albuterol as covariates.
Time Frame: Day 15 (after 2 weeks of treatment)
Population: Participants from the Full Analysis Set, randomized participants who received at least one dose of study drug, who had efficacy data for this outcome measure. Missing data were imputed last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 18.75 µg | Indacaterol 37.5 µg | Indacaterol 75 µg | Indacaterol 150 µg | Salmeterol | Placebo
Number analyzed (Participants) | 82 | 77 | 82 | 80 | 78 | 81
Liters | 2.50 (0.036) | 2.52 (0.037) | 2.59 (0.036) | 2.54 (0.037) | 2.54 (0.037) | 2.42 (0.036)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 1 Day of Treatment
Description: Spirometry was conducted according to internationally accepted standards. The trough FEV1 was defined as the average of the FEV1 measurements taken at 23 hours 10 minutes and 23 hours 45 minutes post dose on day 2. The mixed model used baseline FEV1 and FEV1 prior to and 30 minutes post inhalation of albuterol as covariates.
Time Frame: Day 2 (after 1 day of treatment)
Population: Participants from the Full Analysis Set, randomized participants who received at least one dose of study drug, who had efficacy data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 18.75 µg | Indacaterol 37.5 µg | Indacaterol 75 µg | Indacaterol 150 µg | Salmeterol | Placebo
Number analyzed (Participants) | 83 | 77 | 81 | 82 | 79 | 80
Liters | 2.46 (0.026) | 2.52 (0.027) | 2.54 (0.026) | 2.60 (0.026) | 2.65 (0.027) | 2.45 (0.027)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Safety Population consisting of all participants who received at least one dose of study drug.
Arm/Group | Indacaterol 18.75 µg | Indacaterol 37.5 µg | Indacaterol 75 µg | Indacaterol 150 µg | Salmeterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/81 | 0/84 | 1/85 | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 4/84 | 2/81 | 12/84 | 7/85 | 5/84 | 4/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 18.75 µg (N=84) | Indacaterol 37.5 µg (N=81) | Indacaterol 75 µg (N=84) | Indacaterol 150 µg (N=85) | Salmeterol (N=84) | Placebo (N=84)
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 18.75 µg (N=84) | Indacaterol 37.5 µg (N=81) | Indacaterol 75 µg (N=84) | Indacaterol 150 µg (N=85) | Salmeterol (N=84) | Placebo (N=84)
Headache (Nervous system disorders) | 2 | 2 | 5 | 3 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 8 | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.